CLINICAL TRIAL: NCT04839549
Title: Randomized, Open Label, Prospective Study on the Efficacy and Safety of Dextenza Compared to Topical Fluorometholone in Patients With Ocular Rosacea (ROSE Study)
Brief Title: Efficacy and Safety of Dextenza Compared to Topical Fluorometholone in Patients With Ocular Rosacea
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of patient enrollment
Sponsor: Eye Associates of Central Texas (Other)
Responsible Party: Principal Investigator, Lena Dixit, MD, Principal Investigator, Eye Associates of Central Texas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: The ROSE Study
Record Dates: First submitted 2020-10-19; First posted 2021-04-09 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Ocular Rosacea
MeSH Terms: conditions — Rosacea | interventions — Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dextenza (Intracanalicular ) 0.4mg (Experimental): Dextenza for the treatment of Ocular Rosacea
  Interventions: Drug: Dextenza 0.4Mg Ophthalmic Insert
- Fluoromethalone .01% (Active Comparator): Fluoromethalone .1% BID for 2 weeks then once daily for 2 weeks for the treatment of Ocular Rosacea
  Interventions: Drug: Fluoromethalone .01%

INTERVENTIONS:
Drug: Dextenza 0.4Mg Ophthalmic Insert — Dextenza 0.4Mg Ophthalmic Insert
  Arms: Dextenza (Intracanalicular ) 0.4mg
Drug: Fluoromethalone .01% — Fluoromethalone .01%
  Arms: Fluoromethalone .01%

SUMMARY:
To determine patient preference and treatment outcomes with an intracanalicular dexamethasone (0.4mg) insert compared to a standard steroid drop regimen in the contralateral eye for the treatment of ocular rosacea.

DETAILED DESCRIPTION:
Prospective Open-label Interventional Study Randomized, self-controlled design in which one eye receives Dextenza (Group A) intracanalicular insert and the contralateral eye receives topical fluorometholone 0.1% BID (Group B) for 2 weeks then once daily for 2 weeks for the treatment of ocular rosacea. All patients will be placed on oral doxycycline 100mg BID for one month and tapered to a maintenance dose of 100mg once daily for the remainder of the study. Patient evaluations will be performed at Screening/Baseline, Insertion Day, Month 1 and Month 2.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age, any gender or race
* Provide written informed consent
* Sign the HIPAA form
* Attend all study visits
* Take all study medications as directed
* Be willing to avoid all disallowed medications
* Be willing to avoid all contact lens wear between Dextenza insertion (Visit 2) and Post-op 1 month visit (Visit 3)
* Have a best-corrected visual acuity (BCVA) or greater than or equal to 50 ETDRS letters (20/100 Snellen equivalent) or better in each eye at the screening visit.
* For women of childbearing age (menarche to less than 12 months of menopause who have not undergone surgical sterilization), be willing to have a urine pregnancy test and agree to use a medically acceptable form of birth control throughout the study duration.
* Have a documented diagnosis of Ocular Rosacea and exhibit typical signs or symptoms associated with the diagnosis (irritation, burning, foreign body sensation, redness, itching, inflammation, dry eye, discharge)

Exclusion Criteria:

* Have any allergy or other historical contraindication to the medications in the protocol
* Is unable to use the study medications regularly as directed
* Have any other ocular disease that could affect the subject's ability to participate in the study safely (narrow angle glaucoma, iritis, current infection, elevated intraocular pressure, history of significant steroid response with and IOP >22mmHg, punctal size less than 0.4mm or lid malformation that would preclude insertion of the Dextenza insert)
* Have known history of herpetic eye disease (either active or historical)
* Have a history of refractive surgery within the past 2 years
* Have a history of retinal detachment, diabetic retinopathy, or active retinal disease
* Is currently (within the past 7 days) using an ophthalmic steroid preparation (drop, ointment or insert form)
* Is currently using ocular, topical, or systemic non-steroidal anti-inflammatory drugs (NSAIDs) - Baby aspirin (81mg) is allowed as long as a stable dose has been maintained for at least 30 days prior to Dextenza insertion and will continue to be maintained for the duration of the study
* Have an active infectious disease or is currently taking (or has taken within 7 days of initiation into the study) oral antibiotics
* Is actively being treated with local or systemic immunosuppression, including systemic steroids
* Have a planned ocular or systemic surgery within 30 days of the placement of the Dextenza insert.
* Have used a study drug or participated in a clinical study within 30 days of the beginning of this study
* Is currently pregnant, planning to become pregnant, or breastfeeding
* Is an employee or direct family member of an employee at the clinic site
* Have a diagnosis of any significant uncontrolled illness
* Have a history of alcohol or drug abuse in the past year
* Is a current smoker
* Have used an investigational drug or medical device within 30 days of the study or be concurrently enrolled in another investigational product trial
* Have an intraocular pressure that is less than 5mmHg or greater than 22mmHg or any type of glaucoma
* Is deemed unsafe for the study by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-06 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2022-11-29 (Actual)

PRIMARY OUTCOMES:
Change in OSDI | Accessed at all time points (Day -30 - day -1, week 4, week 8)
  As measured by OSDI questionnaire
Patient preference in treatment therapy | Accessed at Week 4
  As measured by Adapted COMTOL questionnaire

SECONDARY OUTCOMES:
Change in tear breakup time | Accessed at all time points (Day -30 - day -1, week 4, week 8)
  As measured by Fluoroscein (Bioglo strip moistened with saline) placed in the inferior fornix of each eye. A cobalt blue light beam will be used to count the number of seconds between the last blink and the appearance of a dry spot or break in tear film.
Change in Expression of Gland Scale | Accessed at all time points (Day -30 - day -1, week 4, week 8)
  As measured by digitally compressing the lower and upper lids and quantified on a 4-point scale:
  (0- all five glands, 1 - three to four glands, 2 - one to two glands, 3 - zero glands).
  The values will be averaged for each eye.
Change in corneal staining | Accessed at all time points (Day -30 - day -1, week 4, week 8)
  As measured by the NEI/Industry Grading system

IPD SHARING:
Plan to Share IPD: No